CLINICAL TRIAL: NCT03385070
Title: Using Lens Opacities to Predict Salt Sensitivity Hypertension
Brief Title: Salt Sensitivity Hypertension and Lens Opacities
Status: Completed | Type: Observational
Sponsor: Kecioren Education and Training Hospital (Other)
Responsible Party: Principal Investigator, Keçiören Eğitim Araştırma Hastanesi, Cardıologıst, Kecioren Education and Training Hospital
Other Study IDs: 8.3.2017/1325
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Salt Hypertension From Excess Dietary Salt; Lens Opacities
MeSH Terms: conditions — Cataract | interventions — Urinalysis; Blood Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Salt-sensitive group: Patients (n:163)with HT who presented at the emergency service at least once with a minimum increase in their systolic and diastolic blood pressure of 10% after consuming salty foods were included in the SSH group.
  Biomicroscopic lens examination,urine analysis for salt intake estimation,blood pressure measurements
  Interventions: Diagnostic Test: Lens examination
- Salt resistance group: Patients(n:142) who did not exhibit this increase were included in the SRH group
  Biomicroscopic lens examination,urine analysis for salt intake estimation,blood pressure measurements
  Interventions: Diagnostic Test: Lens examination
- Control group: Sex- and age-matched patients(n:124) without a HT diagnosis were included in the control group.
  Biomicroscopic lens examination,urine analysis for salt intake estimation,blood pressure measurements
  Interventions: Diagnostic Test: Lens examination

INTERVENTIONS:
Diagnostic Test: Lens examination — The presence of cortical lens opacity was biomicroscopically examined by two researchers using the diffuse, direct, Scheimpflug and retroillumination from the fundus methods.
  Other Names: urine analysis for salt intake; Blood pressure measurements

SUMMARY:
Salt-sensitive hypertension (SSH) accounts for about the half of all Hypertension (HT) cases .In SSH, Na+/K+-ATPase activity is impaired. Impaired Na+/K+-ATPase activity in the lens epithelium results in cortical opacities in the peripheral equator of the lens.

This study analyzed 305 patients with hypertension aged between 40 and 80 years and 124 non-HT controls. A total of 163 patients with HT who were admitted to the emergency service at least once with a minimum increase of 10% in their systolic and diastolic blood pressure after consuming salted food met the eligible criteria for HT and were included in the SSH group. A total of 142 patients who were previously diagnosed with HT but had no previous history were considered non-SSH. Two researchers examined the presence of cortical lens opacities biomicroscopically using the diffuse, direct, Scheimpflug, and retroillumination from fundus methods.

DETAILED DESCRIPTION:
The number of patients with hypertension (HT) worldwide is estimated to reach 1.56 billion by 2025.HT accounts for almost 50% of deaths due to stroke and coronary artery disease. Salt-sensitive hypertension (SSH) accounts for about the half of all HT cases. Na+ /K+-ATPase activity is impaired in patients with SSH . Impaired Na+ /K+-ATPase activity in the lens epithelium results in cortical opacities in the peripheral equatorial region of the lens.A definite diagnosis of salt sensitivity is difficult, expensive, and associated with low patient compliance. Salt sensitivity is a risk factor for cardiovascular mortality and morbidity regardless of blood pressure and for other diseases such as asthma, gastric carcinoma, osteoporosis, and renal dysfunction. The present study is the first to investigate the potential of using lens opacity to predict SSH.

The transparency of the whole lens is largely based on epithelial cell permeability and Na+ /K+-ATPase activity. Circulation is activated by Na+ /K+-ATPases, which are present at 20-fold normal concentrations, particularly in the equatorial than in the anterior epithelial cells.

The mechanisms associated with SSH pathogenesis, such as signaling pathways involving Src family kinase (SFK), endothelin, connexin, brain natriuretic peptide (BNP), aldosterone, transient receptor protein V4 (TRPV4) ion channel, with-no-lysine kinase-Ste20-like proline/alanine rich kinase/oxidative stress-responsive kinase 1 (WNK-SPAK/OSR1), and Ras-related C3 botulinum toxin substrate (Rac1) , are important to the physiology of the lens epithelium. Compelling studies suggest that inhibition of these pathways may facilitate opacity.

ELIGIBILITY:
Inclusion Criteria:

Salt Sensitivity Hypertension patients Non-SSH, salt-resistant HT (SRH) patients Control patients without HT, aged 40-80 years.

Exclusion Criteria:

Cataracts Diabetes Mellitus Smoking Hypo/hypercalcemia Hyperparathyroidism Eye trauma Coronary artery disease Cardiac failure Renal failure

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The HT and control groups were subdivided into age groups of < 50, 50-59, 60-69, and ≥ 70 years. These age groups comprised 54, 109, 80, and 62 patients in the HT group and 19, 42, 42, and 21 patients in the control group, respectively.
Sampling Method: Probability Sample
Enrollment: 429 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Lens examination | 6 months
  Biomicroscopic lens examination

CONTACTS AND LOCATIONS:
Overall Officials: Şahbender Koç, Cardiologist, Principal Investigator — Keçiören Education and Training Hospital
Locations (1):
- University of Health Sciences.Keçiören Education and Training Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No